CLINICAL TRIAL: NCT07332312
Title: Developing a Culturally Informed Patient Navigation Program to Reduce Delays From Diagnosis to Treatment for Native Americans in a Rural Setting
Brief Title: A Culturally Informed Patient Navigation Program (CFPN) to Reduce Delays Between Diagnosis and Treatment in American Indian and Alaska Native Cancer Patients Living in Rural California
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Cancer Society, Inc. (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 19PS-25-8; NCI-2025-08365 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UP-25-00814; 19PS-25-8 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2025-12-03; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods; Interviews as Topic; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Objective 1 group I (CAB) (Other): Participants serve on a CAB to guide the co-design process of the CFPN program on study.
  Interventions: Other: Discussion
- Objective 1 group II (focus group) (Other): Participants complete a focus group over 1-2 hours in support of the co-design process of the CFPN program on study.
  Interventions: Other: Discussion
- Objective 1 group III (KII) (Other): Participants complete a KII over 30 minutes in support of the co-design process of the CFPN program on study.
  Interventions: Other: Interview
- Objective 2 (CFPN program) (Experimental): Patients engage with the CFPN program navigator as needed and receive a treatment plan based on the patient's needs, goals, and barriers on study. Patients also receive opioid misuse education and care coordination on study.
  Interventions: Other: Educational Intervention; Other: Electronic Health Record Review; Other: Interview; Behavioral: Patient Navigation; Other: Survey Administration; Procedure: Tailored Intervention

INTERVENTIONS:
Other: Discussion — Serve on CAB
  Other Names: Discuss
  Arms: Objective 1 group I (CAB)
Other: Discussion — Complete focus group
  Other Names: Discuss
  Arms: Objective 1 group II (focus group)
Other: Educational Intervention — Receive opioid misuse education and care coordination
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Objective 2 (CFPN program)
Other: Electronic Health Record Review — Ancillary studies
  Arms: Objective 2 (CFPN program)
Other: Interview — Complete KII
  Arms: Objective 1 group III (KII)
Other: Interview — Ancillary studies
  Arms: Objective 2 (CFPN program)
Behavioral: Patient Navigation — Engage with CFPN program navigator
  Other Names: Patient Navigator Program
  Arms: Objective 2 (CFPN program)
Other: Survey Administration — Ancillary studies
  Arms: Objective 2 (CFPN program)
Procedure: Tailored Intervention — Receive treatment plan
  Arms: Objective 2 (CFPN program)

SUMMARY:
This clinical trial develops and tests whether a culturally informed patient navigation program, Community-Focused Patient Navigation (CFPN), works to reduce delays between diagnosis and treatment in American Indian and Alaska Native (AIAN) cancer patients living in rural California. AIAN communities face some of the most severe cancer disparities in the United States, including higher death rates, later-stage diagnoses, and limited access to timely, culturally responsive care. This may be due to barriers such as rural isolation, divided referral systems, or a lack of trust in mainstream healthcare systems. Patient navigation is a care delivery model designed to guide a patient through the healthcare system and address the barriers that prevent patients from accessing timely and effective care. The CFPN program is culturally tailored and designed with AIAN communities in mind. The program provides the patient with a treatment plan based on the patient's unique needs, goals, and barriers. This may be an effective way to reduce delays between diagnosis and treatment in AIAN cancer patients living in rural California.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct a comprehensive community-informed planning process to co-design the Community-Focused Patient Navigation (CFPN) program.

II. Develop and implement an evidence and practice-informed, culturally responsive, CFPN program.

III. Evaluate the implementation and impact of the CFPN program using Practical, Robust Implementation and Sustainability Model (PRISM) and the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) frameworks, along with Indigenous evaluation practices.

OUTLINE: Participants are assigned to 1 of 2 objectives.

OBJECTIVE 1: Participants are assigned to 1 of 3 groups.

GROUP I: Participants serve on a Community Advisory Board (CAB) to guide the co-design process of the CFPN program on study.

GROUP II: Participants complete a focus group over 1-2 hours in support of the co-design process of the CFPN program on study.

GROUP III: Participants complete a key informant interview (KII) over 30 minutes in support of the co-design process of the CFPN program on study.

OBJECTIVE 2:

Patients engage with the CFPN program navigator as needed and receive a treatment plan based on the patient's needs, goals, and barriers on study. Patients also receive opioid misuse education and care coordination on study.

ELIGIBILITY:
Inclusion Criteria:

* CAB: Self-identify as AIAN or have experience working with the AIAN community
* CAB: Are 18 years or older
* CAB: Live within Toiyabe Indian Health Program (TIHP) catchment area(s)
* CAB: Are either a cancer patient/survivor/caregiver and/or a family member of an individual(s) affected by cancer, OR a Board member (ex: Tribal Health Board or Elders Board)
* FOCUS GROUP: Self-identify as AIAN or a family member of an AIAN individual affected by cancer
* FOCUS GROUP: Are 18 years or older
* FOCUS GROUP: Live within TIHP catchment area(s)
* FOCUS GROUP: Are either a cancer patient/survivor/caregiver and/or a family member of an individual(s) affected by cancer, OR a Board member (ex: Tribal Health Board or Elders Board)
* KII: Be a TIHP healthcare staff member
* KII: Be 18 years or older
* KII: Work with AIAN cancer patients in TIHP catchment area
* CFPN PROGRAM IMPLEMENTATION: Have any type of cancer, are in any treatment stage along the cancer continuum
* CFPN PROGRAM IMPLEMENTATION: Self-identify as AIAN or be a TIHP patient
* CFPN PROGRAM IMPLEMENTATION: Live in the TIHP service area
* CFPN PROGRAM IMPLEMENTATION: Receive cancer-related services from TIHP

Exclusion Criteria:

* FOCUS GROUP: Individual with no experience with cancer either as a patient or know someone who is/was a cancer patient at TIHP
* CFPN PROGRAM IMPLEMENTATION: Not a TIHP patient
* CFPN PROGRAM IMPLEMENTATION: Does not currently have cancer or has not previously had cancer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-11-13 (Estimated); Study Completion 2028-11-13 (Estimated)

PRIMARY OUTCOMES:
Focus group themes and emerging codes | Through study completion, up to 2 years
  Will compare themes and emerging codes utilizing qualitative coding computer software. A report will summarize participant responses for each focus group and will be discussed with the Toiyabe Indian Health Program (THIP) co-principal investigator (Co-PI) and staff prior to sharing with the Community Advisory Board (CAB) members.
Key informant interview findings and proposed strategies | Through study completion, up to 2 years
  Will prepare a report with the findings and proposed strategies and discuss it with TIHP Co-PI and CAB.
Qualitative Effectiveness of Community-Focused Patient Navigation (CFPN) program | Through study completion, up to 2 years
  Data collected in interviews focusing on patient's cancer journey and experience with the CFPN program will be analyzed using Dedoose software and an inductive qualitative approach. Two-coder teams will code separately and discuss discrepancies and reconciliations, and the codes will be applied to transcripts and fieldnotes.
Quantitative Effectiveness of Community-Focused Patient Navigation (CFPN) program | Through study completion, up to 2 years
  Using Patient Satisfaction With Cancer Care Scale (Jean-Pierre, 2010) to collect data regarding the effectiveness of the CFPN program. Data will be analyzed using SAS to measure the unilateral satisfaction construct through descriptive statistics (e.g., means, medians, frequencies) and summarizing single-group satisfaction at post-intervention.
Implementation of Community-Focused Patient Navigation (CFPN) program | Through study completion, up to 2 years
  Data will be collected via a study-specific patient survey to examine acceptability, appropriateness, and feasibility of the CFPN program. Data will be analyzed using SAS to calculate means, standard deviations, and ranges.
Attrition | Through study completion, up to 2 years
  Number of patients lost to follow up will be examined to establish the reach of the Community-Focused Patient Navigation (CFPN) program.

CONTACTS AND LOCATIONS:
Overall Officials: Claradina Soto, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Toiyabe Indian Health Project, Bishop, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California